CLINICAL TRIAL: NCT00189956
Title: Phase II, Double-blind, Randomised, Dose-finding Study to Evaluate the Immunogenicity of Three Different Doses of MVA-BN Smallpox Vaccine in 18-30 Year Old Smallpox naïve Healthy Subjects
Brief Title: Dose-finding Study to Evaluate Immunogenicity of Three Different Dose Levels of the IMVAMUNE (MVA-BN) Smallpox Vaccine.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bavarian Nordic (Industry)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: POX-MVA-004
Record Dates: First submitted 2005-09-11; First posted 2005-09-19 (Estimated); Last update posted 2019-01-10 (Actual); Status verified 2018-12

CONDITIONS: Smallpox
MeSH Terms: conditions — Smallpox | interventions — smallpox and monkeypox vaccine modified vaccinia ankara-bavarian nordic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 1 (Active Comparator): healthy, vaccinia naïve subjects 2 x 10E7 TCID50 IMVAMUNE (MVA-BN), subcutaneous
  Interventions: Biological: IMVAMUNE (MVA-BN)
- Group 2 (Active Comparator): healthy, vaccinia naïve subjects 5 x 10E7 TCID50 IMVAMUNE (MVA-BN), subcutaneous
  Interventions: Biological: IMVAMUNE (MVA-BN)
- Group 3 (Active Comparator): healthy, vaccinia naïve subjects
  1 x 10E8 TCID50 IMVAMUNE (MVA-BN), subcutaneous
  Interventions: Biological: IMVAMUNE (MVA-BN)

INTERVENTIONS:
Biological: IMVAMUNE (MVA-BN) — Two vaccinations of 0.5 ml MVA-BN vaccine, separated by a 4 week interval.

SUMMARY:
The objective of the study is to find the optimal dose for the smallpox candidate vaccine IMVAMUNE (MVA-BN). For this purpose the study compares IMVAMUNE (MVA-BN) administered at three different dose levels.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects, aged 18 - 30 years
* Signed informed consent after being advised of the risks and benefits of the study in a language able to understand, and prior to performance of any study specific procedure.
* Free of obvious health problems with acceptable medical history by screening evaluation and physical examination.
* Subject of not of child-bearing potential or all of the following: A urine/serum ß-HCG pregnancy test gives a negative result, use of adequate contraceptive precautions for 30 days before first vaccination.

Exclusion Criteria:

* Known or suspected history of smallpox vaccination or typical vaccinia scar.
* Positive test result in MVA specific ELISA or PRNT at screening.
* Positive result in HIV or HCV antibody test at screening.
* HbsAG positive at screening.
* Pregnancy or breast-feeding.
* Uncontrolled serious infection i.e. not responding to antimicrobial therapy
* History of any serious medical condition, which in the opinion of the investigator, would compromise the safety of the subject.
* History of autoimmune disease
* History of malignancy.
* History of chronic alcohol abuse and/or intravenous drug abuse.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine.
* History of anaphylaxis or severe allergic reaction.
* Acute disease (a moderate or severe illness with or without a fever) at the time of enrolment.
* Any vaccinations within a period starting 30 days prior to administration of the vaccine and ending at study conclusion.
* Chronic administration of immuno-suppressants or other immune-modifying drugs.
* Administration or planned administration of immunoglobulins and/or any blood products during the study period.
* Use of any investigational or non-registered drug or vaccine.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 165 (Actual)
Dates: Start 2003-04; Primary Completion 2003-11 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
ELISA seroconversion rate | Day 42
  Seroconversion rate based on vaccinia-specific Enzyme-linked Immunosorbent Assay (ELISA). Seroconversion is defined as the appearance of antibody titers ≥ detection limit for initially seronegative subjects, or a doubling or more of the antibody titer compared to Baseline titer for initially seropositive subjects. Percentages based on number of subjects with data available.

SECONDARY OUTCOMES:
ELISA seroconversion rate | Days 28, 84
  Seroconversion rate based on vaccinia-specific Enzyme-linked Immunosorbent Assay (ELISA). Seroconversion is defined as the appearance of antibody titers ≥ detection limit for initially seronegative subjects, or a doubling or more of the antibody titer compared to Baseline titer for initially seropositive subjects. Percentages based on number of subjects with data available.
ELISA GMT | Days 28, 42, 84
  Geometric Mean Titers (GMT) based on vaccinia-specific Enzyme-linked Immunosorbent Assay (ELISA). Titers below the detection limit are included with a value of '1'.
PRNT seroconversion rate | Days 28, 42, 84
  Seroconversion rate based on vaccinia-specific Plaque Reduction Neutralization Test (PRNT). Seroconversion is defined as the appearance of antibody titers ≥ detection limit for initially seronegative subjects, or a doubling or more of the antibody titer compared to Baseline titer for initially seropositive subjects. Percentages based on number of subjects with data available.
PRNT GMT | Days 28, 42, 84
  Geometric Mean Titers (GMT) based on vaccinia-specific Plaque Reduction Neutralization Test (PRNT). Titers below the detection limit are included with a value of '1'.
Cytotoxic T-Lymphocyte response | Days 28, 42, 84
  The Cytotoxic T-Lymphocyte (CTL) response was determined by measuring IFNγ producing cells by Intracellular cytokine staining (ICS)
Serious Adverse Events | within 12 weeks
  Incidence, relationship and intensity of any Serious Adverse Event (SAE)
Solicited Local Adverse Events | within 8 days after any vaccination
  Incidence and intensity of solicited local AEs. Percentages based on subjects with at least one completed diary card.
Solicited General Adverse Events | within 8 days after any vaccination
  Incidence of solicited general AEs: Intensity and relationship to vaccination. Percentages based on subjects with at least one completed diary card.
Unsolicited Non-serious Adverse Events | within 31 days after any vaccination
  Occurrence of unsolicited non-serious AEs: Intensity and relationship to vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Rolf Pokorny, M.D., Principal Investigator — Swiss Pharma
Locations (1):
- Swiss Pharma Contract, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] von Krempelhuber A, Vollmar J, Pokorny R, Rapp P, Wulff N, Petzold B, Handley A, Mateo L, Siersbol H, Kollaritsch H, Chaplin P. A randomized, double-blind, dose-finding Phase II study to evaluate immunogenicity and safety of the third generation smallpox vaccine candidate IMVAMUNE. Vaccine. 2010 Feb 3;28(5):1209-16. doi: 10.1016/j.vaccine.2009.11.030. Epub 2009 Nov 25. PMID 19944151